CLINICAL TRIAL: NCT01636011
Title: Effect of Osteopathic Manipulative Medicine on Pulmonary Function and Speech in Parkinson's Disease
Brief Title: Effect of Osteopathic Manipulative Medicine (OMM) on Pulmonary Function and Speech in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BHS-808
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Osteopathic Manipulative Medicine; Speech; Pulmonary Function
MeSH Terms: conditions — Parkinson Disease; Speech

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- OMM Treatment (Experimental): In this group the subjects are given 5 different OMM treatments addressing the thoracic cage.
  Interventions: Other: Osteopathic Manipulative Medicine Treatment
- Light Touch sham (Sham Comparator): In this group the physician uses the dorsum of his hand to the same areas and for the same time that the OMM treatment arm receives.
  Interventions: Other: Light Touch sham

INTERVENTIONS:
Other: Osteopathic Manipulative Medicine Treatment — Osteopathic Manipulative Medicine Treatment
  Arms: OMM Treatment
Other: Light Touch sham — Light Touch sham
  Arms: Light Touch sham

SUMMARY:
The purpose of this study is to investigate the effect of selected Osteopathic Manipulative Medicine (OMM) techniques on the respiratory system of people with Parkinson's Disease (PD) in comparison to light touch. Effectiveness will be measured through pulmonary function tests, chest wall expansion, and voice analysis. Selected subjects will be randomly assigned to one of the two groups: OMM treatment group or light touch group. Although OMM treatment has been used on PD patients, a randomized controlled study has not been done to establish its effect on PD respiratory function. The authors believe that this study will show OMM's effectiveness.

DETAILED DESCRIPTION:
Osteopathic Manipulative Medicine (OMM) on the thoracic cage and diaphragm is commonly used in clinical practice to address myofascial imbalances, including muscle spasms to improve thoracic cage excursion. Prior research has demonstrated that manual approaches applied to the thoracic cage have positive results with lung function and reducing inflammation.

Parkinson's disease (PD) is a common disabling and progressive neuro-degenerative disorder. Morbidity and mortality are frequently associated with pulmonary dysfunction in patients with PD. Pulmonary function tests (PFT) have been utilized to document respiratory impairment in PD patients. Researchers estimate that 89% of people with PD have speech and voice disorders including disorders of laryngeal, respiratory and articulatory function.

These authors hypothesize that performing OMM on the thoracic cage of PD subjects will show improvement in PFT, chest expansion, and speech production. Subjects with PD meeting the criteria for the study will be randomly assigned to either an OMM treatment or light touch control group. Each subject will be involved in one treatment visit. During this visit, the following will be measured before and after OMM or light touch procedures: maximal and minimal chest circumference; sound pressure, duration, and perceptual measures during sustained vowel phonation and Rainbow Reading; Forced Vital Capacity (FVC), Forced Expiratory Volume/1 second (FEV1), Peak Expiratory Flow (PEF), Forced Expiratory Flow 25%-75% (FEF25-75%), and Maximal Voluntary Ventilation (MVV). Data analysis will be performed with SPSS using Analysis of Covariance to measure significance.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with Parkinson's Disease
* on a stable medication dose
* over the age of 18

Exclusion Criteria:

* no clinical diagnosis of Parkinson's Disease
* - medication that might cause pulmonary dysfunction
* inability to perform PFT because of anatomical abnormalities
* clinical signs of dementia
* pacemaker that interferes with pectoral traction
* metastatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function tests | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Yao, DO, Principal Investigator — NYIT
Locations (1):
- NYIT NYCOM Academic Health Care Center, Old Westbury, New York, United States

REFERENCES:
- [Background] Degenhardt BF, Kuchera ML. Update on osteopathic medical concepts and the lymphatic system. J Am Osteopath Assoc. 1996 Feb;96(2):97-100. doi: 10.7556/jaoa.1996.96.2.97. PMID 8838905
- [Background] Belcastro MR, Backes CR, Chila AG. Bronchiolitis: a pilot study of osteopathic manipulative treatment, bronchodilators, and other therapy. J Am Osteopath Assoc. 1984 May;83(9):672-6. No abstract available. PMID 6725033
- [Background] Sleszynski SL, Kelso AF. Comparison of thoracic manipulation with incentive spirometry in preventing postoperative atelectasis. J Am Osteopath Assoc. 1993 Aug;93(8):834-8, 843-5. PMID 8407387
- [Background] Sathyaprabha TN, Kapavarapu PK, Pall PK, Thennarasu K, Raju TR. Pulmonary functions in Parkinson's disease. Indian J Chest Dis Allied Sci. 2005 Oct-Dec;47(4):251-7. PMID 16255396
- [Background] Yamada H, Murahashi M, Takahashi H, Kai K, Shibuya S, Jimi T, Wakayama Y, Yamada M. [Respiratory function impairment in patients with Parkinson's disease--a consideration on the possible pathogenetic relation to autonomic dysfunction]. Rinsho Shinkeigaku. 2000 Feb;40(2):125-30. Japanese. PMID 10835931
- [Background] Polatli M, Akyol A, Cildag O, Bayulkem K. Pulmonary function tests in Parkinson's disease. Eur J Neurol. 2001 Jul;8(4):341-5. doi: 10.1046/j.1468-1331.2001.00253.x. PMID 11422431
- [Background] Ramig LO, Sapir S, Fox C, Countryman S. Changes in vocal loudness following intensive voice treatment (LSVT) in individuals with Parkinson's disease: a comparison with untreated patients and normal age-matched controls. Mov Disord. 2001 Jan;16(1):79-83. doi: 10.1002/1531-8257(200101)16:13.0.co;2-h. PMID 11215597
- [Background] Goetz CG, Poewe W, Rascol O, Sampaio C, Stebbins GT, Counsell C, Giladi N, Holloway RG, Moore CG, Wenning GK, Yahr MD, Seidl L; Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. Movement Disorder Society Task Force report on the Hoehn and Yahr staging scale: status and recommendations. Mov Disord. 2004 Sep;19(9):1020-8. doi: 10.1002/mds.20213. PMID 15372591
- [Background] Rapaport MH, Schettler P, Breese C. A preliminary study of the effects of a single session of Swedish massage on hypothalamic-pituitary-adrenal and immune function in normal individuals. J Altern Complement Med. 2010 Oct;16(10):1079-88. doi: 10.1089/acm.2009.0634. PMID 20809811
- [Background] Bockenhauer SE, Chen H, Julliard KN, Weedon J. Measuring thoracic excursion: reliability of the cloth tape measure technique. J Am Osteopath Assoc. 2007 May;107(5):191-6. PMID 17596587